CLINICAL TRIAL: NCT00194415
Title: A Randomized Clinical Trial of Antenatal vs Delayed (Post Partum) Testing for HSV Type-Specific Antibodies Among Pregnant Women.
Brief Title: A Study of HSV Testing Among Pregnant Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An interim data analysis found no significant difference between testing groups.
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Anna Wald, MD, MPH / Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-9950-E/A; P01AI030731 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Herpes Simplex; Pregnancy
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): HSV-2 antepartum testing
  Interventions: Procedure: Type specific serologic HSV testing
- 2 (Other): Subjects will receive safer-sex counseling during pregnancy
  Interventions: Behavioral: Safer-sex counseling

INTERVENTIONS:
Behavioral: Safer-sex counseling — Subjects will receive safer-sex counseling during pregnancy
  Arms: 2
Procedure: Type specific serologic HSV testing — Subjects will be testing for HSV by Western Blot
  Arms: 1

SUMMARY:
The objective of the study is to evaluate the acceptance and effect of type- specific HSV serologic testing of pregnant women on sexual behavior at the end of pregnancy.

DETAILED DESCRIPTION:
The study hypothesis is that women with antepartum testing who are identified as susceptible to HSV-1 or HSV-2 will have reduced unprotected coital activity and reduced unprotected oral-genital activity compared to those who did not receive antepartum testing. The objective of the study is to evaluate the acceptance, and effect of type-specific HSV serologic testing of pregnant women on sexual behavior at the end of pregnancy.

Upon enrollment, study participants will be randomized into either of two type-specific HSV serologic testing and counseling regimens:

* Group 1: Antepartum and postpartum testing. Subjects will be made aware of their antepartum testing results.
* Group 2: Antepartum blood draw and postpartum testing. Subjects' specimens will be tested at the same time.

Women in group 2 will receive information about herpes infection and how to decrease their chance of acquiring infection during pregnancy. Subjects will be asked to keep a diary of sexual activity and return to the clinic every 4 weeks until delivery.

ELIGIBILITY:
Inclusion Criteria:

* 14 years of age or older
* Pregnant less than 28 weeks at time of enrollment
* No previous HSV serology within the past year
* able to comprehend english

Exclusion Criteria:

* History of genital herpes
* HIV seropositive
* Any contraindication for sexual activity during pregnancy

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2004-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The reduction of unprotected coital or oral-genital activity in women who are identified as being susceptible to HSV-1 or HSV-2. | From time of enrollment (pregnant less than 28 weeks at the time of enrollment) to delivery

SECONDARY OUTCOMES:
To determine HSV seroconversion rates in Group 1 versus Group 2 | From time of enrollment (pregnant less than 28 weeks at the time of enrollment) to delivery
To determine rates of neonatal HSV infection in Groups 1 & 2. | From time of enrollment (pregnant less than 28 weeks at the time of enrollment) to delivery
To determine viral shedding characteristics in those mother-infant pairs where seroconversion occurs. | From time of enrollment (pregnant less than 28 weeks at the time of enrollment) to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Money, MD, Principal Investigator — University of British Columbia; Anna Wald, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada